CLINICAL TRIAL: NCT06849427
Title: Effects of Multicomponent Exercise on Quality of Life, Coping With Stress, and Well-Being in Older Women: A Randomized Controlled Trial
Brief Title: Effects of Multicomponent Exercise on Quality of Life, Coping With Stress, and Well-Being in Older Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-002
Record Dates: First submitted 2025-01-14; First posted 2025-02-27 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-02

CONDITIONS: Quality of Life; Coping; Well-being; Older People; Woman's Health; Exercise
Keywords: quality of life; coping; well being; older people; exercise; women's health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 20 experimental, 20 control
Who Masked: Participant
Masking Description: 20 control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Multi-component exercise application will be performed
  Interventions: Other: multicomponent exercise intervention
- Control group (No Intervention): Multi-component exercise will not be applied

INTERVENTIONS:
Other: multicomponent exercise intervention — Multicomponent Exercise Program
  A. Flexibility B. Targeted Strength Training C. Balance and Mobility
  1. Center of Gravity Control Training
  2. Multisensory Training
  3. Postural Strategy Training
  4. Gait Pattern Development Variation Training
  5. Dual Task Exercises . D. Cardiovespiratory Fitness
  Arms: Exercise group

SUMMARY:
The aim of this study is to evaluate the effects of multi-component exercise on quality of life, coping with stress and well-being in elderly women.

The objectives of the study are;

* To determine the contribution of multi-component exercise to active and healthy aging in elderly women
* To present the effects of multi-component exercise on quality of life, coping with stress and well-being in elderly women and to create data to guide practitioners for nursing care practices.

This study will determine whether multi-component exercise will make a positive contribution to quality of life, well-being and coping strategies in elderly women and will contribute to the deepening of existing knowledge on the effects of multi-component exercise on health.

DETAILED DESCRIPTION:
Aging is a natural and inevitable process of change that begins in the fetal period and continues until death in all living things. Old age refers to a period in which many people experience feelings of loss, lose their physical, functional, psychological and social independence and increase their dependency. The World Health Organization (WHO) accepts the age limit as 65 years and above, while the United Nations accepts it as 60 years and above. In parallel with the developments in technology, science and health, 9.3% of the world's population and 9.1% in our country constitute the elderly population. 61% of the population aged 80 and above in the world are women, and the female/male ratio in this population is increasing day by day.

Biological differences cause women to spend more than a third of their lives in old age and to have more health-seeking behaviors due to men's higher rates of smoking, alcohol and substance use. This situation causes older women to experience chronic diseases, violence, abuse and reproductive health problems, psychological and mental problems, care and housing problems longer than older men. According to the study of Ko et al. (2019), it was found that women have lower socioeconomic and health status than men, and their health status and social service needs are higher than men. In addition, studies have shown that urinary incontinence, osteoporosis, vision, hearing problems, cardiovascular diseases such as hypertension, which are common in elderly women, negatively affect their mobility and quality of life.

The care that should be given to the elderly should be multifaceted, and in addition to physical and medical aspects, social and psychological aspects should not be neglected. Functional losses and social losses that occur in old age naturally affect women more. Coping with stress is defined as a series of cognitive and behavioral efforts aimed at managing special needs that exceed the individual's internal resources. Although the life behaviors developed by women to cope with stress in the literature vary from culture to culture, most studies have focused on education, physical activity/exercise, healthy nutrition, stress management, developing healthy behaviors, and preventing diseases and osteoporosis. Some problems such as increasing health problems in old age, loss of professional and social status, loss of function, and increased dependence on others deteriorate the quality of life and negatively affect well-being. Although wellness is simply defined as a process, a lifestyle, it consists of multifaceted sub-dimensions such as social, physical, and spiritual well-being. In geriatric studies aimed at maintaining well-being, studies are carried out on social activities, psychological support, and exercise, nutrition, and the ability of the individual to continue their daily activities independently. In the study of Östh et al. (2019), it is reported that yoga is effective in improving well-being, mobility, mood and cognition, and that yoga can be added to the exercise program of the elderly. In addition, in the study of Sorusa et al., it was determined that yoga applied during the climacteric period positively affects the quality of life and well-being.

Current geriatric studies target active aging and report that exercise is necessary for a healthy aging process. While exercising increases muscle mass, muscle strength, balance and speed, it also helps elderly individuals increase their independence and reduce functional disability. WHO's exercise recommendations for elderly individuals include both strength exercises and balance exercises to reduce the risk of falls, as well as aerobic exercises. The recommendation for older adults is 150 minutes of moderate-intensity exercise per week, and it is stated that it is more appropriate to divide this time into certain days of the week. Epidemiological studies have shown that people with high levels of physical activity have lower levels of depression and anxiety. On the other hand, high levels of habitual physical activity are associated with a reduced risk of cognitive decline, dementia, and Alzheimer's disease in later life. Physical exercise improves memory function in older people with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Being a woman over 60
* Agreeing to participate in the research
* Being able to speak and understand Turkish

Exclusion Criteria:

* Those who have previously engaged in active regular exercise and continue to do so
* Those who are unable to do physical exercise due to any illness
* Those who are involved in another study simultaneously with this study outside of routine practices
* Those who have another neurological or psychiatric diagnosis affecting their cognitive status

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Assesment | pre-intervention and immediately after the intervention
  The World Health Organization Quality of Life Scale Short Form is a 26-question shortened version of the 100-question World Health Organization Quality of Life Assesment (WHOQOL) scale, which was prepared to assess how an individual perceives their quality of life. The scale, which includes closed-ended questions, consists of four sub-domains: physical, social, environmental, and psychological. The physical domain consists of questions 3, 4, 10, 15, 16, 17, and 18; the psychological domain consists of questions 5, 6, 7, 11, 19, and 26; the social domain consists of questions 20, 21, 22; and the environmental domain consists of questions 8, 9, 12, 13, 14, 23, 24, and 25. The scale does not have a full score, and an increase in score indicates an improvement in quality of life. The Turkish validity and reliability study of the scale was conducted by Eser and his colleagues in 1999, and during their work, a national question was added to the scale, increasing the number of questions to 2

SECONDARY OUTCOMES:
Stress Coping Style Scale | pre-intervention and immediately after the intervention
  The scale, developed by Folkman and Lazarus in 1988, was adapted to Turkish by Şahin and Durak in 1995 and its validity and reliability studies were conducted. Later, Şahin and Durak (1995) adapted the Ways of Coping with Stress Scale for university students. The scale consists of 30 items and is a 4-point Likert type (0=not at all appropriate, 1=not appropriate, 2=appropriate, 3=completely appropriate). Only items 1 and 9 are scored in reverse. The scale, which has two dimensions, consists of five subsections. The first of its dimensions is aimed at effectively solving the encountered problem and is called "Problem-oriented/active" and consists of the subsections "Applying to social support", "Optimistic approach" and "Self-confident approach". The other dimension is related to emotional coping, which is considered as ineffective coping, and is called "Emotion-oriented/passive" and consists of the subsections "Helpless approach" and "Submissive approach". Individuals who can effectiv

OTHER OUTCOMES:
Well-Being Scale | pre-intervention and immediately after the intervention
  The Turkish adaptation of the Well-Being Scale, developed by Diener et al. (2009), was conducted by Fidan and Usta. The scale has a 7-point Likert structure. The highest score that can be obtained from the scale is 56, and the lowest score is 8. There are no reverse-scored items in the scale. High scores obtained from the scale indicate that the relevant individual has a high level of well-being. It was conducted by Fidan and Usta (2013) on a total of 385 high school 4th grade students, 166 (%43) girls and 219 (%57) boys. The Cronbach alpha internal consistency coefficient of the Well-Being Scale was found to be .83.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Antalya Aktif Yaşlı Merkezi, Konyaalti, Antalya
  - Antalya Aktif Yaşlı Merkezi, Antalya

IPD SHARING:
Plan to Share IPD: Yes
Participants' demographic data and scale scores will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: February 2025-February 2026
Access Criteria: The data obtained in the study will be analyzed using the free trial version of SPSS Statistics (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistics (number, percentage, mean, standard deviation) will be used when evaluating the data. The normality test will be decided according to the significance value of the "Shapiro-Wilk" test. As a result of the normality test, the "Mann-Whitney U test" will be used for analyzes related to scales that do not show normal distribution, and the "Wilcoxon W" test will be used to analyze pre-test-post-test mean scores. In analyzes related to scales that show normal distribution, the "Independent Samples t test" and the "Paired Samples t test" will be used to analyze pre-test-post-test mean scores. "Reliability Analysis" will be performed in calculating the "Cronbach alpha" coefficients of the scales. In the study, p values under 0.05 will be considered significant.

REFERENCES:
- [Result] Muchiri WA, Olutende OM, Kweyu IW, Vurigwa E. Meaning of Physical Activities for the Elderly: A Review. Am J Sports Sci Med 2018;6:79-83. https://www.researchgate.net/publication/327602163_Meaning_of_Physical_Activities_for_the_Elderly_A_Review
- [Result] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Result] Ko KY, Kwok ZCM, Chan HY. Effects of yoga on physical and psychological health among community-dwelling older adults: A systematic review and meta-analysis. Int J Older People Nurs. 2023 Sep;18(5):e12562. doi: 10.1111/opn.12562. Epub 2023 Aug 14. PMID 37577926
- [Result] Varela S, Ayan C, Cancela JM, Martin V. Effects of two different intensities of aerobic exercise on elderly people with mild cognitive impairment: a randomized pilot study. Clin Rehabil. 2012 May;26(5):442-50. doi: 10.1177/0269215511425835. Epub 2011 Nov 24. PMID 22116953
- See also: Effects of two different intensities of aerobic exercise on elderly people with mild cognitive impairment: a randomized pilot study — https://pubmed.ncbi.nlm.nih.gov/22116953/
- Available data/document: Individual Participant Data Set: sibelcynk@gmail.com — https://www.antalya.edu.tr/tr — If online access is not available: instructions for how to obtain information